CLINICAL TRIAL: NCT00782132
Title: Access to Infertility Services in Ontario for Couples in Which One or Both Partners is HIV-Positive
Brief Title: Access to Infertility Services: Clinic Perspective
Status: Completed | Type: Observational
Sponsor: Unity Health Toronto (Other)
Responsible Party: Sponsor
Other Study IDs: 06-248
Record Dates: First submitted 2008-10-29; First posted 2008-10-31 (Estimated); Last update posted 2023-12-12 (Actual); Status verified 2023-12

CONDITIONS: Infertility
Keywords: Infertility Services, HIV, pregnancy planning
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

SUMMARY:
Since the identification of the human immunodeficiency virus (HIV) and the acquired immunodeficiency syndrome (AIDS) in the 1980s, there have been significant advances made in the management and long-term prognosis for infected individuals. Currently, with the advent of highly active antiretroviral therapy (HAART), HIV-positive individuals may live a healthy and productive life for years to decades after diagnosis. As life expectancy has increased, this group of people has begun to engage in family planning. This has created a need for access to advanced reproductive technologies and fertility treatments. While attempting to achieve pregnancy, utilization of these services can help to minimize the risk of transmission in serodiscordant couples, and can allow treatment of subfertile couples. Access to these services may be limited in Ontario for a variety of reasons. The purpose of this study is to determine the access to infertility clinics and services in Ontario for couples in which one or both partners is infected with HIV.

ELIGIBILITY:
Inclusion Criteria:

* All Ontario clinics offering advanced reproductive/infertility services

Exclusion Criteria:

* none

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Ontario clinics offering advanced reproductive/infertility services
Sampling Method: Non-Probability Sample
Enrollment: 23 (Actual)
Dates: Start 2006-11; Primary Completion 2008-05 (Actual); Study Completion 2008-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mona Loutfy, MD, Principal Investigator — Women's College Research Institute
Locations (1):
- St. Michael's Hospital, Toronto, Ontario, Canada

REFERENCES:
- [Derived] Yudin MH, Shapiro HM, Loutfy MR. Access to infertility services in Canada for HIV-positive individuals and couples: a cross-sectional study. Reprod Health. 2010 May 12;7:7. doi: 10.1186/1742-4755-7-7. PMID 20462451